CLINICAL TRIAL: NCT05021562
Title: Zedula Special Drug Use Observational Study "Ovarian Cancer"
Brief Title: A Study of Niraparib in Patients With Ovarian Cancer in Clinical Practice
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Niraparib-4001; jRCT2031210289 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-08-24; First posted 2021-08-25 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Niraparib 200-300 milligrams (mg): Arm description: Niraparib 200 mg, capsules, orally, once daily. For adult participants weighing 77 kilograms (kg) or more and with platelet count 150,000/mcrL or higher before the first dose of this drug, niraparib 300 mg, capsules, orally, once daily.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib capsules

SUMMARY:
The main aim of this study is to check for side effects from treatment with niraparib.

The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

During the study, participants with ovarian cancer will take capsules of niraparib (Zedula) once a day according to their clinic's standard practice. The study doctors will check for side effects from niraparib for 1 year after treatment starts.

ELIGIBILITY:
Inclusion Criteria:

An individual who corresponds to any of the following:

* Ovarian cancer patients after initial chemotherapy (maintenance therapy)
* Patients with platinum antineoplastic drug sensitive recurrent ovarian cancer (maintenance therapy)
* Recurrent ovarian cancer with platinum-sensitive homologous recombination repair defects.

Exclusion Criteria:

Has a history of hypersensitivity to any of the ingredients of this drug.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An individual who corresponds to any of the following: ovarian cancer patients after initial chemotherapy (maintenance therapy), patients with platinum antineoplastic drug sensitive recurrent ovarian cancer (maintenance therapy), or recurrent ovarian cancer with platinum-sensitive homologous recombination repair defects.
Sampling Method: Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Event of Myelosuppression | 1 year
  An Adverse Event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product. It does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with AE of myelosuppression will be reported.
Number of Participants with Adverse Event of Hypertension | 1 year
  Number of participants with AE of hypertension will be reported.
Number of Participants with Adverse Event of Posterior Reversible Encephalopathy Syndrome | 1 year
  Number of participants with AE of posterior reversible encephalopathy syndrome will be reported.
Number of Participants with Adverse Event of Interstitial Lung Disease | 1 year
  Number of participants with AE of interstitial lung disease will be reported.
Number of Participants with Adverse Event of Secondary Malignant Tumors | 1 year
  Number of participants with AE of secondary malignant tumors will be reported.
Number of Participants with Adverse Event of Thromboembolism | 1 year
  Number of participants with AE of thromboembolism will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve or Maintain Any Best Overall Response Category in Population of Recurrent Ovarian Cancer Participants with Platinum-Sensitive Homologous Recombination Repair Defects | 1 year
  Percentage of participants who achieve or maintain any best overall response category best overall response in population of recurrent ovarian cancer participants with platinum-sensitive homologous recombination repair defects will be reported. Best overall response will be assessed with reference to the excerpts from Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Best overall response is defined as the level of best response in assessment with complete response (CR), partial response (PR), progressive disease (PD), stable disease (SD) and not evaluable (NE) during the observational period.
Number of Participants who Experienced Exacerbation Assessed by Investigator during the Study | 1 year
  Exacerbation is defined as death or worsened symptom or disease assessed by investigator through tumor assessments, tumor marker assessments, and clinical assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/613700d1c61629002b6311e2